CLINICAL TRIAL: NCT03339713
Title: A Randomized, Double-blind, Placebo-controlled Phase 2a Study to Evaluate the Safety and Immunogenicity of Seasonal Influenza Vaccine and Ad26.RSV.preF, With and Without Co-administration, in Adults Aged 60 Years and Older in Stable Health
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Seasonal Influenza Vaccine and an Adenovirus Serotype 26- Based Vaccine Encoding for the Respiratory Syncytial Virus Pre-fusion F Protein (Ad26.RSV.preF), With and Without Co-administration, in Adults Aged 60 Years and Older in Stable Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108403; VAC18193RSV2003 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ad26.RSV.preF Plus Fluarix Then Placebo: Group 1 (Experimental): Participants will receive intramuscular injection of 1*10^11 viral particles (vp) of an adenovirus serotype 26- based vaccine encoding for the respiratory syncytial virus pre-fusion F protein (Ad26.RSV.preF) on 1 arm administered at the same time as a commercially available seasonal influenza vaccine (Fluarix) on the other arm at Day 1, and intramuscular injection of placebo on Day 29.
  Interventions: Biological: Ad26.RSV.preF; Biological: Fluarix; Biological: Placebo
- Placebo Plus Fluarix Then Ad26.RSV.preF: Group 2 (Experimental): Participants will receive intramuscular injection of placebo administered at the same time as a commercially available seasonal influenza vaccine (Fluarix) on Day 1, and 1*10^11 vp of Ad26.RSV.preF on Day 29.
  Interventions: Biological: Ad26.RSV.preF; Biological: Fluarix; Biological: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.preF — Ad26.RSV.preF will be administered as intramuscular injection at a dose of 1*10^11 vp.
  Other Names: JNJ-64400141
Biological: Fluarix — Fluarix will be administered as intramuscular injection.
Biological: Placebo — Placebo will be administered as intramuscular injection of sterile 0.9 percent (%) saline for injection.

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of the concomitant administration of an adenovirus serotype 26- based vaccine encoding for the respiratory syncytial virus pre-fusion F protein (Ad26.RSV.preF) and seasonal influenza vaccine versus the administration of seasonal influenza vaccine alone in terms of humoral immune response expressed by the geometric mean titers (GMTs) of hemagglutination inhibition (HI) antibody titers against all four influenza vaccine strains 28 days after the administration of influenza vaccine, and to assess the safety and tolerability of a single dose of 1*10^11 viral particles (vp) of Ad26.RSV.preF, administered intramuscularly to participants aged greater than or equal to 60 years separately or concomitantly with seasonal influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, is willing to participate in the study and attend all scheduled visits, and is willing and able to comply with all study procedures and adhere to the prohibitions and restrictions specified in this protocol
* Before randomization, a woman must be:

  1. Postmenopausal (A postmenopausal state is defined as no menses for 12 months without an alternative medical cause) and
  2. Not intending to conceive by any methods
* In the investigator's clinical judgment, participant must be either in good or stable health, and not at risk of serious complications from influenza. Participants may have underlying illnesses such as hypertension, type 2 diabetes, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms/signs are medically controlled. If they are on medication for a condition, the medication dose must have been stable for at least 12 weeks (or only small, clinically non-significant changes have been made in the judgement of the Principal Investigator) preceding vaccination and expected to remain stable for the duration of the study. Participants will be included on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed on Day 1
* From the time of first vaccination through 3 months after the second dose of study vaccine, participant agrees not to donate blood
* Participant must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has acute illness (this does not include minor illnesses such as diarrhea) or temperature greater than or equal to (>=) 38.0 degree Celsius (ºC) within 24 hours prior to the first dose of study vaccine; enrollment at a later date is permitted
* Participant has a serious chronic disorder, including severe chronic obstructive pulmonary disease or clinically significant congestive heart failure, requirement for supplemental oxygen, end stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has had major surgery (per the investigator's judgment), within 4 weeks before dosing, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 6 months after the final dose of study vaccine
* Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Coastal Carolina Research Center, Mt. Pleasant, South Carolina, United States

REFERENCES:
- [Derived] Sadoff J, De Paepe E, Haazen W, Omoruyi E, Bastian AR, Comeaux C, Heijnen E, Strout C, Schuitemaker H, Callendret B. Safety and Immunogenicity of the Ad26.RSV.preF Investigational Vaccine Coadministered With an Influenza Vaccine in Older Adults. J Infect Dis. 2021 Feb 24;223(4):699-708. doi: 10.1093/infdis/jiaa409. PMID 32851411

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo: Participants received a single dose of intramuscular injection of 1*10^11 viral particles (vp) of Adenovirus serotype 26 Respiratory Syncytial Virus pre-fusion conformation stabilized F protein (Ad26.RSV.preF) on Day 1 along with Fluarix administered at the same time, followed by placebo as second vaccine on Day 29.
- Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp): Participants received a single dose of intramuscular injection of placebo on Day 1 along with Fluarix administered at the same time, followed by 1*10^11 vp Ad26.RSV.preF as second vaccine on Day 29.
Period: Overall Study
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Started | 90 | 90
Completed | 86 | 88
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp) | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Median (Full Range); unit: years] | 64 [60 to 82] | 66 [60 to 81] | 65 [60 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 33 | 34 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 89 | 89 | 178
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 79 | 81 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Antibody Titers as Measured by Hemagglutination Inhibition Assay (HAI) Against Each of the Four Vaccine Influenza Strains
Description: Humoral immune responses expressed by the geometric mean titers (GMTs) of HI antibody titers against each of four influenza vaccine strains (A/Michigan, A/Hong Kong, B/Brisbane and B/Phuket). Serum specimens were tested for the presence of HAI antibodies to influenza vaccine strains. The HAI assay was conducted using serum samples from participants.
Time Frame: 28 days after vaccination (Day 29)
Population: The Per-protocol influenza immunogenicity (PPII) set included participants who were randomized and received the first vaccination for whom immunogenicity data are available, excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 85 | 89
Titers
  A/Michigan strain | 215 [160 to 289] | 168 [125 to 226]
  A/Hong Kong strain | 98 [73 to 131] | 80 [61 to 103]
  B/Brisbane strain | 39 [31 to 49] | 40 [31 to 51]
  B/Phuket strain | 35 [28 to 43] | 35 [27 to 46]
Statistical Analysis 1: Comparison: Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo vs Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp); A/Michigan strain: Based on Welch-Satterthwaite t-interval method. The difference (Group 2 minus Group 1) and CI in log-transformed HI antibody titers were calculated for each of the 4 influenza vaccine strains, and were back-transformed (by exponentiation) to a GMT ratio (Group 2 / Group 1) and the corresponding CI; Test type: Non-Inferiority — Non-inferiority of Group 2 versus Group 1 in terms of the HI antibody titers against all four influenza vaccine strains 28 days after the administration of influenza vaccine, using a non-inferiority margin of 2 for the GMT ratio (Group 2 / Group 1); p < .001, t-test, 1 sided; Geometric Mean Ratio = 0.8, 90% CI 2-sided [0.55 to 1.11]
Statistical Analysis 2: Comparison: Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo vs Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp); A/Hong Kong strain: Based on Welch-Satterthwaite t-interval method. The difference (Group 2 minus Group 1) and CI in log-transformed HI antibody titers were calculated for each of the 4 influenza vaccine strains, and were back-transformed (by exponentiation) to a GMT ratio (Group 2 / Group 1) and the corresponding CI; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < .001, t-test, 1 sided; Geometric Mean Ratio = 0.8, 90% CI 2-sided [0.59 to 1.12]
Statistical Analysis 3: Comparison: Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo vs Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp); B/Brisbane strain: Based on Welch-Satterthwaite t-interval method. The difference (Group 2 minus Group 1) and CI in log-transformed HI antibody titers were calculated for each of the 4 influenza vaccine strains, and were back-transformed (by exponentiation) to a GMT ratio (Group 2 / Group 1) and the corresponding CI; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < .001, t-test, 1 sided; Geometric Mean Ratio = 1.0, 90% CI 2-sided [0.77 to 1.34]
Statistical Analysis 4: Comparison: Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo vs Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp); B/Phuket strain: Based on Welch-Satterthwaite t-interval method. The difference (Group 2 minus Group 1) and CI in log-transformed HI antibody titers were calculated for each of the 4 influenza vaccine strains, and were back-transformed (by exponentiation) to a GMT ratio (Group 2 / Group 1) and the corresponding CI; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < .001, t-test, 1 sided; Geometric Mean Ratio = 1.0, 90% CI 2-sided [0.76 to 1.36]

2. Primary Outcome: Post-dose 1: Percentage of Participants Reporting at Least 1 Solicited Local and Systemic Adverse Events (AEs)
Description: Percentage of participants reporting at least 1 solicited local and systemic AEs were shown. Solicited local AEs: erythema, swelling/induration, and pain/tenderness. Solicited systemic AEs: fatigue, headache, myalgia, arthralgia, chills, nausea and fever. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product.
Time Frame: Up to 7 days post-dose 1 on Day 1 (Day 8)
Population: The Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26.RSV.preF or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 90 | 90
Percentage of participants
  Post-dose 1: Solicited local AEs | 80.0 | 45.6
  Post-dose 1: Solicited systemic AEs | 63.3 | 27.8

3. Primary Outcome: Post-dose 2: Percentage of Participants Reporting at Least 1 Solicited Local and Systemic AEs
Description: as for outcome 2
Time Frame: Up to 7 days post-dose 2 on Day 29 (Day 36)
Population: The Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26.RSV.preF or placebo). Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 88 | 90
Percentage of participants
  Post-dose 2: Solicited local AEs | 6.8 | 76.7
  Post-dose 2: Solicited systemic AEs | 18.2 | 70.0

4. Primary Outcome: Post-dose 1: Percentage of Participants With Unsolicited AEs
Description: Percentage of participants with unsolicited AEs were shown. Unsolicited AEs are all AEs for which participants were specifically not questioned in the participant diary. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product.
Time Frame: Up to 28 days post-dose 1 on Day 1 (Day 29)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 90 | 90
Percentage of participants | 36.7 | 33.3

5. Primary Outcome: Post-dose 2: Percentage of Participants With Unsolicited AEs
Description: Percentage of participants with unsolicited AEs 2 were shown. Unsolicited AEs are all AEs for which participants were specifically not questioned in the participant diary. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product.
Time Frame: Up to 28 days post-dose 2 on Day 29 (Day 57)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 88 | 90
Percentage of participants | 18.2 | 18.9

6. Primary Outcome: Post-dose 1: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 6 months post-dose 1 (Day 183)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 90 | 90
Percentage of participants | 0 | 0

7. Primary Outcome: Post-dose 2: Percentage of Participants With SAEs
Description: as for outcome 6
Time Frame: Up to 6 months post-dose 2 (Day 211)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 88 | 90
Percentage of participants | 1 | 1

8. Secondary Outcome: Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers
Description: RSV A2 neutralizing titers of the vaccine-induced immune response was assessed through virus neutralization assay.
Time Frame: Baseline and Day 29 (post Ad26.RSV.preF)
Population: The Per-protocol RSV Immunogenicity (PPRI) set included all randomized and fully vaccinated participants (all three vaccinations, ie, Fluarix Quadrivalent, Ad26.RSV.preF and placebo) for whom immunogenicity data are available, excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here 'n' (number analyzed) included all participants who were analyzed at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 88 | 90
Titers
  Baseline | 497 [429 to 576] | 539 [458 to 636]
  Day 29: number analyzed (Participants) | 88 | 86
  Day 29 | 1404 [1208 to 1633] | 1690 [1433 to 1993]

9. Secondary Outcome: RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)- Pre-Fusion
Description: GMT (ELISA units per litre [EU/L]) of RSV F protein in pre-fusion form by ELISA was reported.
Time Frame: Baseline and Day 29 (post Ad26.RSV.preF)
Population: The PPRI set included all randomized and fully vaccinated participants (all three vaccinations, ie, Fluarix Quadrivalent, Ad26.RSV.preF and placebo) for whom immunogenicity data are available, excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. Here 'n' (number analyzed) included all evaluable participants who were analyzed at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 88 | 90
EU/L
  Baseline | 333 [289 to 384] | 315 [267 to 371]
  Day 29: number analyzed (Participants) | 88 | 86
  Day 29 | 781 [694 to 879] | 814 [711 to 932]

10. Secondary Outcome: RSV Fusion Protein (F-protein) GMTs as Assessed by ELISA- Post-Fusion
Description: GMT (EU/L) to RSV F protein in post-fusion form by ELISA was reported.
Time Frame: Baseline and Day 29 (post Ad26.RSV.preF)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Group 1: Ad26.RSV.preF (1*10^11 vp) Plus Fluarix Then Placebo | Group 2: Placebo Plus Fluarix Then Ad26.RSV.preF (1*10^11 vp)
Number analyzed (Participants) | 88 | 90
EU/L
  Baseline | 256 [223 to 295] | 236 [203 to 274]
  Day 29: number analyzed (Participants) | 88 | 86
  Day 29 | 506 [444 to 577] | 484 [426 to 549]

ADVERSE EVENTS:
Time Frame: SAEs were collected up to end of study (Day 211) and non-serious AEs were collected up to 28 days Post-dose 1 (Day 29) and Post-dose 2 (Day 57).
Description: The Full Analysis Set (FAS) included all participants who were randomized and received at least one dose of study vaccine, regardless of the occurrence of protocol deviations and vaccine type (Fluarix Quadrivalent, Ad26.RSV.preF or placebo). Reported AEs were presented as pre-specified in the study protocol.
Groups:
- Group 1 Post-Dose 1: Ad26.RSV.preF (1*10^11 vp) + Fluarix Quadrivalent (Day 1): Participants received a single dose of intramuscular injection of 1*10^11 vp (viral particles) of Ad26.RSV.preF on Day 1 along with Fluarix administered at the same time.
- Group 2 Post-Dose 1: Placebo + Fluarix Quadrivalent (Day 1): Participants received a single dose of intramuscular injection of matching placebo on Day 1 along with Fluarix administered at the same time.
- Group 1 Post-Dose 2: Placebo (Day 29): Participants received a single dose of intramuscular injection of matching placebo on Day 29.
- Group 2 Post-Dose 2: Ad26.RSV.preF (Day 29): Participants received a single dose of intramuscular injection of Ad26.RSV.preF on Day 29.
Arm/Group | Group 1 Post-Dose 1: Ad26.RSV.preF (1*10^11 vp) + Fluarix Quadrivalent (Day 1) | Group 2 Post-Dose 1: Placebo + Fluarix Quadrivalent (Day 1) | Group 1 Post-Dose 2: Placebo (Day 29) | Group 2 Post-Dose 2: Ad26.RSV.preF (Day 29)
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90 | 0/88 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 1/88 | 1/90
Other Adverse Events (participants affected / at risk) | 22/90 | 18/90 | 13/88 | 14/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Post-Dose 1: Ad26.RSV.preF (1*10^11 vp) + Fluarix Quadrivalent (Day 1) (N=90) | Group 2 Post-Dose 1: Placebo + Fluarix Quadrivalent (Day 1) (N=90) | Group 1 Post-Dose 2: Placebo (Day 29) (N=88) | Group 2 Post-Dose 2: Ad26.RSV.preF (Day 29) (N=90)
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Renal Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertensive Emergency (Vascular disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Post-Dose 1: Ad26.RSV.preF (1*10^11 vp) + Fluarix Quadrivalent (Day 1) (N=90) | Group 2 Post-Dose 1: Placebo + Fluarix Quadrivalent (Day 1) (N=90) | Group 1 Post-Dose 2: Placebo (Day 29) (N=88) | Group 2 Post-Dose 2: Ad26.RSV.preF (Day 29) (N=90)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Injection Site Pruritus (General disorders) | 1 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 10 | 11 | 7 | 5
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Blood Pressure Increased (Investigations) | 5 | 4 | 3 | 5
Headache (Nervous system disorders) | 2 | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Although qualification of the site was satisfactory for peripheral blood mononuclear cells (PBMC) processing,during the study PBMC processing resulted in much lower yield than expected, which have affected the quality of PBMC. While sample quality requirements on sample viability were met for most samples,viability was considered lower than commonly expected.An indication of possible suboptimal quality of PBMC samples were also be a low baseline responses observed in comparison to other studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03339713/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT03339713/SAP_001.pdf